CLINICAL TRIAL: NCT01359488
Title: A Blinded Placebo Controlled Single Ascending Dose Phase 1 for Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics After Subcutaneous Administration of VRS-317 in Adults With Growth Hormone Deficiency
Brief Title: VRS-317 in Adult Subjects With Growth Hormone Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Versartis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VRS-317 1a
Record Dates: First submitted 2011-05-13; First posted 2011-05-24 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth Hormone Deficiency; rhGH; hGH; Versartis; AGHD; Hormones; Hormone substitute; Endocrin System disease; Bone disease; Bone disease, developmental; Bone diseases; Musculoskeletal diseases; Bone diseases, endocrine; Metabolism diseases; Hypopituitarism; Pituitary disease; Hypothalmic disease; Brain disease; Growth Hormone Releasing Hormone; Hormone replacement therapy; IGF-I; IGFBP-3
MeSH Terms: conditions — Dwarfism, Pituitary; Bone Diseases; Bone Diseases, Developmental; Musculoskeletal Diseases; Bone Diseases, Endocrine; Hypopituitarism; Pituitary Diseases; Brain Diseases | interventions — Insulin-Like Growth Factor I; Insulin-Like Growth Factor Binding Protein 3; Hormones; Hormones, Hormone Substitutes, and Hormone Antagonists; Growth and Development; National Institute of Arthritis and Musculoskeletal and Skin Diseases (U.S.); Hormone Replacement Therapy; Growth Hormone-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- VRS-317 Safety Arm 1 (Experimental): VRS-317 Single injection SC of dose level 1 (based on 90 kg patient)
  Placebo Single SC injection Dose Volume matched to active treatment volume
  Interventions: Drug: VRS-317
- VRS-317 Safety Arm 2 (Experimental): VRS-317 Single injection SC of dose level 2 (based on 90 kg patient)
  Placebo Single SC injection Dose Volume matched to active treatment volume
  Interventions: Drug: VRS-317
- VRS-317 Safety Arm 3 (Experimental): VRS-317 Single injection SC of dose level 3 (based on 90 kg patient)
  Placebo Single SC injection Dose Volume matched to active treatment volume
  Interventions: Drug: VRS-317
- VRS-317 Safety Arm 4 (Experimental): VRS-317 Two injections SC of dose level 4 (based on 90 kg patient)
  Placebo Two SC injection Dose matched to treatment volume
  Interventions: Drug: VRS-317
- VRS-317 Safety Arm 5 (Experimental): VRS-317 Two injections SC of dose level 5 (based on 90 kg patient)
  Placebo Two SC injections Dose Volume matched to active treatment volume
  Interventions: Drug: VRS-317

INTERVENTIONS:
Drug: VRS-317 — VRS-317 Single Dose
  Other Names: Growth Hormone Deficiency; rhGH; hGH; AGHD; IGF-I; IGFBP-3; Hormones; Hormone Substitutes; Endocrine System Disease; Bone Diseases; Bone Diseases, Developmental; Musculoskeletal Diseases; Bone Disease, Endocrine; Metabolic Diseases; Hypopituitarism; Pituitary Disease; Hypothalmic Disease; Growth Hormone Replacement Therapy; Hormone Replacement Therapy; Growth Hormone Releasing Hormone; Versartis; VRS317
  Arms: VRS-317 Safety Arm 1
Drug: VRS-317 — VRS-317 Single Dose
  Other Names: Growth Hormone Deficiency; rhGH; hGH; AGHD; IGF-I; IGFBP-3; Hormones; Hormone Substitutes; Endocrine System Disease; Bone Diseases; Bone Diseases, Developmental; Musculoskeletal Diseases; Bone Disease, Endocrine; Metabolic Diseases; Hypopituitarism; Pituitary Disease; Hypothalmic Disease; Growth Hormone Replacement Therapy; Hormone Replacement Therapy; Growth Hormone Releasing Hormone; Versartis; VRS317
  Arms: VRS-317 Safety Arm 2
Drug: VRS-317 — VRS-317 Single Dose
  Other Names: Growth Hormone Deficiency; rhGH; hGH; AGHD; IGF-I; IGFBP-3; Hormones; Hormone Substitutes; Endocrine System Disease; Bone Diseases; Bone Diseases, Developmental; Musculoskeletal Diseases; Bone Disease, Endocrine; Metabolic Diseases; Hypopituitarism; Pituitary Disease; Hypothalmic Disease; Growth Hormone Replacement Therapy; Hormone Replacement Therapy; Growth Hormone Releasing Hormone; Versartis; VRS317
  Arms: VRS-317 Safety Arm 3
Drug: VRS-317 — VRS-317 Single dose
  Other Names: Arms:; Other Names:; Growth Hormone Deficiency; rhGH; hGH; AGHD; IGF-I; IGFBP-3; Hormones; Hormone Substitutes; Endocrine System Disease; Bone Diseases; Bone Diseases, Developmental; Musculoskeletal Diseases; Bone Disease, Endocrine; Metabolic Diseases; Hypopituitarism; Pituitary Disease; Hypothalmic Disease; Growth Hormone Replacement Therapy; Hormone Replacement Therapy; Growth Hormone Releasing Hormone; Versartis
  Arms: VRS-317 Safety Arm 4
Drug: VRS-317 — VRS-317 Single dose
  Other Names: Growth Hormone Deficiency; rhGH; hGH; AGHD; IGF-I; IGFBP-3; Hormones; Hormone Substitutes; Endocrine System Disease; Bone Diseases; Bone Diseases, Developmental; Musculoskeletal Diseases; Bone Disease, Endocrine; Metabolic Diseases; Hypopituitarism; Pituitary Disease; Hypothalmic Disease; Growth Hormone Replacement Therapy; Hormone Replacement Therapy; Growth Hormone Releasing Hormone; Versartis; VRS317
  Arms: VRS-317 Safety Arm 5

SUMMARY:
The purpose of this research study is to determine the safety and tolerability of up to five doses of VRS-317 in Adult Growth Hormone Deficient patients.

* Patients will be evaluated for evidence of activity of VRS-317 by measurement of changes from baseline in insulin-like growth factor-1 (IGF-I) and binding protein (IGFBP-3), and bone turnover (bone alkaline phosphatase)
* Descriptive pharmacokinetic (PK) and pharmacodynamic (PD) parameters (IGF-I and IGFBP-3) will be determined by standard model independent methods based on the plasma concentration-time data of each subject. These parameters include: Cmax, Tmax, AUCavg, AUC0-inf, and t1/2.
* The purpose is to determine the appropriate dose of VRS-317 to maintain a normal range (for appropriate age/gender) for IGF-I levels in adult patients for up to one month after administration of a single dose

DETAILED DESCRIPTION:
The study is a placebo controlled single ascending dose (SAD) study in adult GHD patients currently receiving daily rhGH therapy. After screening patients are withdrawn from daily rhGH therapy for a minimum of 7 days (maximum of 60 days) prior to randomization for treatment. Patients will be randomised within a treatment group that is currently being enrolled once the patient has passed the pre-dose screening criteria.

Documented confirmation (medical history) of GHD during adulthood by a minimum of one or more GH stimulation tests is required such as:

* insulin tolerance test (ITT; peak hGH ≤ 5.0 ng/mL),
* arginine alone (peak hGH ≤ 0.4 ng/mL);
* arginine + growth-hormone-releasing hormone* (see below);
* or glucagon stimulation test (peak hGH ≤ 3.0 ng/mL) OR
* at least 3 other pituitary hormone deficiencies and a low IGF-I for age/gender appropriate normal range

Each patient will be randomised to receive either the investigational product, VRS-317 (Cohorts A-E), or placebo (Cohort F) in a 4:1 ratio.

Subjects will be monitored for safety throughout their participation in the study. To ensure patient safety, two patients (1 active, 1 placebo) in the first treatment group, one from Cohort A and one from Cohort F1, will be dosed in a blinded manner and monitored for 48 hr prior to dosing the remaining 8 patients. The 8 remaining patients will be blinded and randomized to the first treatment group. Vital signs, clinical lab values, adverse events (AEs) and concomitant medications (CMs) will be captured. AEs will be graded using the Common Terminology Criteria for Adverse Events (CTCAE v 4.0)1, and the Primary Dermal Irritation Scoring Scale; AEs will be coded using the MedDRA2 dictionary and CMs using the WHO Drug dictionary. Prior to escalating to a higher dose level, safety data will be reviewed by the principal investigator (PI), co-PIs, the Sponsor, and the medical monitor for any potential safety risk to subjects.

Patients will participate for a total of 83-215 days. A 7-60 day withdrawal phase (no daily rhGH therapy) is followed by receiving assigned doses on Day 1 of Treatment Phase, PK/PD and safety assessments for 30 days, and an additional 30 days of follow up.

Safety evaulations will be performed to assess safety including but not limited to:

* Physical examination
* Vital signs (including sitting/supine blood pressure)
* Laboratory tests: hematology, chemistry, urinalysis, and pregnancy testing (in women of child-bearing age)
* Adverse events and concomitant medications
* Glucose metabolism: Fasting and post-prandial plasma glucose and fasting insulin pre-study and at pre-scheduled timepoints during the study (per Assessment Table)
* Lipid profile will be assessed pre-study and at pre-scheduled timepoints during the study (per Assessment Table)
* Assessment for adrenal insufficiency prior to enrollment and at Day 30 (not performed on patients with documented history of adrenal insufficiency)
* Evaluation of injection site reactions
* Anti-VRS-317 antibody assay (pre-dose, Day 30 (end of study) and Day 60) last follow up visit
* Safety monitoring will continue for up to 60 days post-dose

ELIGIBILITY:
Inclusion Criteria:

1. Age 25 to 65 years
2. Negative serum pregnancy test for females of childbearing potential
3. Documented confirmation (medical history) of GHD during adulthood by one or more GH stimulation test
4. If taking hormone replacement therapy other than rhGH, patient must be on a stable course of treatment for 2 months prior to enrollment
5. Pituitary disorder associated with GHD has been clinically stable for at least 6 months
6. Currently receiving daily recombinant human growth hormone (rhGH) injections for treatment of GHD for a minimum of 28 days
7. Willing and able to give informed consent
8. Within one year from enrollment, normal result from screening including: mammogram (women), pap smear (women over 25), Men over 50 years old: digital rectal exam

Exclusion Criteria:

1. Subjects who have received systemic treatment for any bacterial, viral or fungal infection within 30 days of the first study drug dosing (prophylactic acyclovir for HSV is permitted)
2. Subjects with documented history of diabetes mellitus or inadequate glucose control as defined by fasting plasma glucose level of greater than 126 mg/dL (7 mM) or HbA1c of ≥ 6.5% at screening
3. Subjects with untreated adrenal insufficiency.
4. Free thyroxine below normal reference range or TSH above normal reference range
5. Current use of oral or inhaled steroids except for physiological maintenance doses of oral glucocorticoids in patients with multiple pituitary hormone deficiencies
6. Women using oral estrogens, including birth control pills, during study (transdermal estrogen patches are allowed)
7. Current significant cardiovascular, cerebrovascular, pulmonary, neurological (not related to GHD), renal or hepatobillary disease
8. Presence of retinopathy or papillaedema
9. Documented history of persistent (unresolved without medical intervention) or recurring migraines, edema, arthralgia (not related to osteoarthritis), or nausea
10. History of drug or alcohol abuse.
11. Must not have documented prior history of HIV, HBV or HCV infection(testing not required)
12. Prior history of cancer excluding adequately treated non-melanoma skin cancers or adequately treated in situ carcinoma of the cervix
13. Women who are pregnant or breastfeeding
14. Unwilling to use two effective birth control methods until Day 60 of Treatment Phase
15. Pre-existing antibodies to human growth hormone at time of screening (screening samples must be below pre-specified cut-off for positive anti-hGH antibody titer)
16. Treatment with an investigational drug within past 30 days prior to screening
17. Unable to comply with requirements of this study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of single dose of VRS-317 | 30 days
  This study will evaluate the differences between VRS-317 dose levels and placebo for adverse events. Summaries will be provided for each dose cohort and for the combined dose cohorts including the number of patients with adverse events. All subjects who receive at least one dose of VRS-317 or placebo will be included in the safety analysis. Summaries of all adverse events (AEs)and serious adverse events (SAEs)will be classified according to severity and relationship to study drug.

SECONDARY OUTCOMES:
Determine the pharmacokinetic (PK) profile of VRS-317 administered SC | 30 days
  Parameters
  * Pharmacokinetic (PK)parameters are determined from WinNonLin analysis using a one compartment model. [Timeframe = 30 days] Cmax Tmax AUCavg AUC0-inf t1/2
  * Parmacodynamic (PD)parameters are determined from WinNonLin analysis using a one compartment model. [Timeframe = 30 days] Cmax Tmax AUCavg AUC0-inf t1/2
  * IGF-I and IGFBP-3 values compared against baseline parameters and parameters obtained from daily rhGH treatment. [Timeframe = 90 days]

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kipnes, MD, Principal Investigator — Diabetes and Glandular Disease Clinic
Locations (1):
- Diabetes and Glandular Disease Clinic, San Antonio, Texas, United States

REFERENCES:
- [Derived] Yuen KC, Conway GS, Popovic V, Merriam GR, Bailey T, Hamrahian AH, Biller BM, Kipnes M, Moore JA, Humphriss E, Bright GM, Cleland JL. A long-acting human growth hormone with delayed clearance (VRS-317): results of a double-blind, placebo-controlled, single ascending dose study in growth hormone-deficient adults. J Clin Endocrinol Metab. 2013 Jun;98(6):2595-603. doi: 10.1210/jc.2013-1437. Epub 2013 Apr 12. PMID 23585663